CLINICAL TRIAL: NCT01482377
Title: Phase Ia/Ib, Open-Label, Multicenter, Dose-Escalation Study Followed by an Extension Phase to Evaluate the Safety, Pharmacokinetics and Activity of RO5479599, A Glycoengineered Antibody Against HER3, Administered Either Alone (Part A) or in Combination With Cetuximab (Part B) or in Combination With Erlotinib (Part C) in Patients With Metastatic and/or Locally Advanced Malignant HER3-Positive Solid Tumors of Epithelial Cell Origin
Brief Title: A Study of RO5479599 Alone or in Combination With Cetuximab or Erlotinib in Participants With Metastatic and/or Locally Advanced Malignant Human Epidermal Growth Factor Receptor (HER3) Expressing Solid Tumors of Epithelial Cell Origin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP27771; 2011-002698-53 (EudraCT Number)
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — lumretuzumab; Cetuximab; Erlotinib Hydrochloride

ARMS (4):
- Part A: RO5479599 Dose Escalation (Experimental): Participants will receive a dose of 100 milligrams (mg) RO5479599 followed by dose escalation from Day 1 of Cycle 1. RO5479599 dose will be escalated as monotherapy in approximately 6 cohorts with dose increments between cohorts of up to 100 percent (%) until MTD.
  Interventions: Drug: RO5479599
- Part B: RO5479599 Dose Escalation + Cetuximab (Experimental): Participants will receive RO5479599 in combination with cetuximab. Escalation of RO5479599 in combination with cetuximab will start in a standard 3+3 design until MTD/OBD is reached. If the initial combination is not tolerated, further cohorts will be dosed with the same dose of cetuximab and lower doses of RO5479599.
  Interventions: Drug: RO5479599; Drug: Cetuximab
- Part C: RO5479599 Dose Escalation + Erlotinib (Experimental): Participants will receive RO5479599 in combination with erlotinib. Escalation of RO5479599 in combination with erlotinib will start in a standard 3+3 design until MTD/OBD is reached. If the initial combination is not tolerated, further cohorts will be dosed with the same dose of erlotinib and lower doses of RO5479599.
  Interventions: Drug: RO5479599; Drug: Erlotinib
- Imaging (IMG) Substudy (Experimental): RO5479599 will be administered with zirconium- 89-labeled RO5479599.
  Interventions: Drug: RO5479599; Drug: zirconium-89-labeled RO5479599

INTERVENTIONS:
Drug: RO5479599 — RO5479599 will be administered Q2W or Q3W (other regimen could be explored based on observations during dose escalation part).
Drug: Cetuximab — Cetuximab will be administered via intravenous (IV) infusion at a starting dose of 400 mg/m^2 for the first infusion, followed by doses of 250 mg/m^2 for subsequent infusions.
  Arms: Part B: RO5479599 Dose Escalation + Cetuximab
Drug: Erlotinib — Erlotinib, at a dose of 150 mg will be administered.
  Arms: Part C: RO5479599 Dose Escalation + Erlotinib
Drug: zirconium-89-labeled RO5479599 — Single dose of radiolabeled drug will be administered.
  Arms: Imaging (IMG) Substudy

SUMMARY:
This dose-escalating study consists of 3 parts (A, B and C) and will evaluate the safety, pharmacokinetics and efficacy of RO5479599, alone or in combination with cetuximab or erlotinib, in participants with metastatic and/or locally advanced malignant HER3-positive solid tumors. Cohorts of participants will receive escalating doses of intravenous RO5479599 as monotherapy (Part A) or in combination with cetuximab (in Part B) or with erlotinib (in Part C) followed by an extension phase for each part.

In an imaging substudy, participants will receive one or two doses of zirconium-89-labeled RO5479599 (89ZrRO5479599) in addition to unlabeled RO5479599 to evaluate the in vivo biodistribution and organ pharmacokinetics of RO5479599.

ELIGIBILITY:
Inclusion Criteria:

All Parts (A, B and C)

* European Cooperative Oncology Group (ECOG) performance status 0-2
* Histologically confirmed metastatic and/or locally advanced malignant HER3-expressing solid tumors of epithelial origin
* Availability of tissue and willingness to perform fresh pretreatment biopsies
* Participants for whom no standard therapy exists
* All acute toxic effects of any prior radiotherapy, chemotherapy or surgical procedure must have resolved to Grade less than or equal to (</= 1), except for alopecia and Grade 2 peripheral neuropathy
* Adequate hematological, renal and liver function
* Participants with Gilbert's syndrome will be eligible for the study

Part B extension cohort: In addition to the above inclusion criteria, participants will be eligible if they have metastatic and/or locally advanced non-small cell lung cancer or squamous cell carcinoma of the head and neck or colorectal cancer (wild type with positive epidermal growth factor receptor [EGFR] expression)

Part C extension cohort: In addition to the above inclusion criteria, participants will be eligible only if they have metastatic and/or locally advanced squamous non-small cell lung cancer

Exclusion Criteria:

* Known or clinically suspected central nervous system (CNS) primary tumors or metastases including leptomeningeal metastases. History or clinical evidence of CNS metastases unless they have been previously treated, are asymptomatic and have had no requirement for steroids or enzyme-inducing anticonvulsants in the last 14 days
* Evidence of significant uncontrolled concomitant diseases or disorders
* Active or uncontrolled infections
* Known Human immuno deficiency virus (HIV) infection
* Therapy with antibody or immunotherapy concurrently or within 14 days prior to first dose of study drug
* Regular immunosuppressive therapy
* Concurrent high dose of systemic corticosteroids (greater than (>) 20 milligrams per day [mg/day] dexamethasone or equivalent for > 7 consecutive days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2011-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events | Baseline up to 28 days after last dose (approximately 48 months)
Maximum Tolerated Dose (MTD) or Optimal Biological Dose (OBD) of RO5479599 | Cycle 1 Day 1 (cycle length = 14 or 21 days) up to 28 days
Number of Participants With Dose Limiting Toxicities (DLTs) | Cycle 1 Day 1 (cycle length = 14 or 21 days) up to 28 days
Standardized Uptake Value (SUV) of 89ZrRO5479599 Determined by Positron Emission Tomography (PET) Scan Over Regions of Interest (ROI) | From baseline to Day 8

SECONDARY OUTCOMES:
Percentage Change From Baseline in Standardized Uptake Value (SUV) of 89ZrRO5479599 at Pharmacodynamic (PD) active dose as Determined by PET Scan | From baseline to Day 22
Part A: Recommended Phase II Dose (RPTD) of RO5479599 in Monotherapy | Cycle 1 Day 1 (cycle length = 14 or 21 days) up to 28 days
Part B: Recommended Phase II Dose of RO5479599 in Combination With Cetuximab | Cycle 1 Day 1 (cycle length = 14 or 21 days) up to 28 days
Part C: Recommended Phase II Dose of RO5479599 in Combination With Erlotinib | Cycle 1 Day 1 (cycle length = 14 or 21 days) up to 28 days
Percentage of Participants With Objective Response According to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | From screening to disease progression, death, withdrawal, or end of study (assessed at screening, then every eighth week for two weekly schedule [Q2W] and every ninth week for three weekly schedule [Q3W] up to approximately 48 months)
Percentage of Participants With Disease Control According to RECIST version 1.1 | From screening to disease progression, death, withdrawal, or end of study (assessed at screening, then every eighth week for Q2W and every ninth week for Q3W up to approximately 48 months)
Duration of Response According to RECIST version 1.1 | From screening to disease progression, death, withdrawal, or end of study (assessed at screening, then every eighth week for Q2W and every ninth week for Q3W up to approximately 48 months)
Progression Free Survival According to RECIST version 1.1 | From screening to disease progression, death, withdrawal, or end of study (assessed at screening, then every eighth week for Q2W and every ninth week for Q3W up to approximately 48 months)
Maximum Serum Concentration (Cmax) of RO5479599 for Q2W Schedule | Pre-infusion (PrI, 0 hours [hr]) & end of infusion (EOI, 1.5 hr) on each 2-week cycle (Cy); 2, 5 hr post-infusion (PoI) on Cy1 Day 1 (D1), Cy1 Days 2, 3, 5, 8, 12; 2 hr PoI on Cy4D1; Cy4 Days 2, 3, 5, 8; Cy8 Days 2, 5, 8 (up to 48 months overall)
Cmax of RO5479599 for Q3W Schedule | PrI (0 hr) & EOI (1.5 hr) on each 3-week Cy; 3 hr PoI on Cy1 D1, Cy1 Days 2, 4, 8, 12, 14, 19, 21; 3 hr PoI on Cy4 D1, Cy8 D1; Days 2, 4, 8, 12, 14, 19, 21 on Cy4 and Cy8 (up to 48 months overall)
Trough Serum Concentration (Cmin) for Q2W Schedule | PreI (0 hr) on D1 of each cycle from Cy2 (up to 48 months overall) (Cycle length = 14 days)
Cmin for Q3W Schedule | PreI (0 hr) on D1 of each cycle from Cy2 (up to 48 months overall) (Cycle length = 21 days)
Time to Reach Maximum Serum Concentration (Tmax) of RO5479599 for Q2W Schedule | PrI (0 hr) & EOI (1.5 hr) on each 2-week Cy; 2, 5 hr PoI on Cy1 D1, Cy1 Days 2, 3, 5, 8, 12; 2 hr PoI on Cy4D1; Cy4 Days 2, 3, 5, 8; Cy8 Days 2, 5, 8 (up to 48 months overall)
Tmax of RO5479599 for Q3W Schedule | PrI (0 hr) & EOI (1.5 hr) on each 3-week Cy; 3 hr PoI on Cy1 D1, Cy1 Days 2, 4, 8, 12, 14, 19, 21; 3 hr PoI on Cy4 D1, Cy8 D1; Days 2, 4, 8, 12, 14, 19, 21 on Cy4 and Cy8 (up to 48 months overall)
Area Under the Plasma Concentration-Time Curve (AUC) of RO5479599 for Q2W Schedule | PrI (0 hr) & EOI (1.5 hr) on each 2-week Cy; 2, 5 hr PoI on Cy1 D1, Cy1 Days 2, 3, 5, 8, 12; 2 hr PoI on Cy4D1; Cy4 Days 2, 3, 5, 8; Cy8 Days 2, 5, 8 (up to 48 months overall)
AUC of RO5479599 for Q3W Schedule | PrI (0 hr) & EOI (1.5 hr) on each 3-week Cy; 3 hr PoI on Cy1 D1, Cy1 Days 2, 4, 8, 12, 14, 19, 21; 3 hr PoI on Cy4 D1, Cy8 D1; Days 2, 4, 8, 12, 14, 19, 21 on Cy4 and Cy8 (up to 48 months overall)
Clearance (CL) of RO5479599 for Q2W Schedule | PrI (0 hr) & EOI (1.5 hr) on each 2-week Cy; 2, 5 hr PoI on Cy1 D1, Cy1 Days 2, 3, 5, 8, 12; 2 hr PoI on Cy4D1; Cy4 Days 2, 3, 5, 8; Cy8 Days 2, 5, 8 (up to 48 months overall)
CL of RO5479599 for Q3W Schedule | PrI (0 hr) & EOI (1.5 hr) on each 3-week Cy; 3 hr PoI on Cy1 D1, Cy1 Days 2, 4, 8, 12, 14, 19, 21; 3 hr PoI on Cy4 D1, Cy8 D1; Days 2, 4, 8, 12, 14, 19, 21 on Cy4 and Cy8 (up to 48 months overall)
Volume of Distribution (Vd) of RO5479599 for Q2W Schedule | PrI (0 hr) & EOI (1.5 hr) on each 2-week Cy; 2, 5 hr PoI on Cy1 D1, Cy1 Days 2, 3, 5, 8, 12; 2 hr PoI on Cy4D1; Cy4 Days 2, 3, 5, 8; Cy8 Days 2, 5, 8 (up to 48 months overall)
Vd of RO5479599 for Q3W Schedule | PrI (0 hr) & EOI (1.5 hr) on each 3-week Cy; 3 hr PoI on Cy1 D1, Cy1 Days 2, 4, 8, 12, 14, 19, 21; 3 hr PoI on Cy4 D1, Cy8 D1; Days 2, 4, 8, 12, 14, 19, 21 on Cy4 and Cy8 (up to 48 months overall)
Accumulation Ratio of RO5479599 for Q2W Schedule | PrI (0 hr) & EOI (1.5 hr) on each 2-week Cy; 2, 5 hr PoI on Cy1 D1, Cy1 Days 2, 3, 5, 8, 12; 2 hr PoI on Cy4D1; Cy4 Days 2, 3, 5, 8; Cy8 Days 2, 5, 8 (up to 48 months overall)
Accumulation Ratio of RO5479599 for Q3W Schedule | PrI (0 hr) & EOI (1.5 hr) on each 3-week Cy; 3 hr PoI on Cy1 D1, Cy1 Days 2, 4, 8, 12, 14, 19, 21; 3 hr PoI on Cy4 D1, Cy8 D1; Days 2, 4, 8, 12, 14, 19, 21 on Cy4 and Cy8 (up to 48 months overall)
Terminal Elimination Half-Life (t1/2) of RO5479599 for Q2W Schedule | PrI (0 hr) & EOI (1.5 hr) on each 2-week Cy; 2, 5 hr PoI on Cy1 D1, Cy1 Days 2, 3, 5, 8, 12; 2 hr PoI on Cy4D1; Cy4 Days 2, 3, 5, 8; Cy8 Days 2, 5, 8 (up to 48 months overall)
t1/2 of RO5479599 for Q3W Schedule | PrI (0 hr) & EOI (1.5 hr) on each 3-week Cy; 3 hr PoI on Cy1 D1, Cy1 Days 2, 4, 8, 12, 14, 19, 21; 3 hr PoI on Cy4 D1, Cy8 D1; Days 2, 4, 8, 12, 14, 19, 21 on Cy4 and Cy8 (up to 48 months overall)
Serum Concentration of RO5479599 at Time of Tumor Progression (Cprog) for Q2W Schedule | PrI (0 hr) & EOI (1.5 hr) on each 2-week Cy; 2, 5 hr PoI on Cy1 D1, Cy1 Days 2, 3, 5, 8, 12; 2 hr PoI on Cy4D1; Cy4 Days 2, 3, 5, 8; Cy8 Days 2, 5, 8 (up to 48 months overall)
Cprog of RO5479599 for Q3W Schedule | PrI (0 hr) & EOI (1.5 hr) on each 3-week Cy; 3 hr PoI on Cy1 D1, Cy1 Days 2, 4, 8, 12, 14, 19, 21; 3 hr PoI on Cy4 D1, Cy8 D1; Days 2, 4, 8, 12, 14, 19, 21 on Cy4 and Cy8 (up to 48 months overall)
Serum Concentration of RO5479599 at the Time of Tumor Response for Q2W Schedule | At the time of objective response (up to 48 months)
Serum Concentration of RO5479599 at the Time of Tumor Response for Q3W Schedule | At the time of objective response (up to 48 months)
Serum Concentration of RO5479599 at the Time of DLT for Q2W Schedule | At the time of DLT (up to 28 days)
Serum Concentration of RO5479599 at the Time of DLT for Q3W Schedule | At the time of DLT (up to 28 days)
Serum Concentration of RO5479599 at the Time of Tumor and Skin Biopsy (Cb) for Q2W Schedule | PrI (0 hr) on Cy1D1 and on Cy1 Day 14 (Cycle length = 14 days)
Cb of RO5479599 for Q3W Schedule | PrI (0 hr) on Cy1D1 and on Cy1 Day 21 (Cycle length = 21 days)
Serum Concentration of RO5479599 at the Time of PET Scan (Cpet) for Q2W Schedule | PrI (0 hr) on Cy1D1, Cy1 Day 14, and Cy4 Day 14 (Cycle length = 14 days)
Cpet of RO5479599 for Q3W Schedule | PrI (0 hr) on Cy1D1, Cy1 Day 21, and Cy3 Day 21 (Cycle length = 21 days)
Serum Concentration of RO5479599 at Time of Infusion-Related Reactions (IRRs) for Q2W Schedule | At the time of IRR (up to 48 months)
Serum Concentration of RO5479599 at Time of IRRs for Q3W Schedule | At the time of IRR (up to 48 months)
Change from Baseline in T Lymphocytes Cell Count for Q2W Schedule | PrI (0 hr) on Cy1D1 (Baseline), Cy1 Day 14, and Cy4 Day 14 (Cycle length = 14 days)
Change from Baseline in T lymphocytes Cell Count for Q3W Schedule | PrI (0 hr) on Cy1D1 (Baseline), Cy1 Day 21, and Cy3 Day 21 (Cycle length = 21 days)
Change from Baseline in Natural Killer Cell Count for Q2W Schedule | PrI (0 hr) on Cy1D1 (Baseline), Cy1 Day 14, and Cy4 Day 14 (Cycle length = 14 days)
Change from Baseline in Natural Killer Cell Count for Q3W Schedule | PrI (0 hr) on Cy1D1 (Baseline), Cy1 Day 21, and Cy3 Day 21 (Cycle length = 21 days)
Change from Baseline in Macrophages Cell Count for Q2W Schedule | PrI (0 hr) on Cy1D1 (Baseline), Cy1 Day 14, and Cy4 Day 14 (Cycle length = 14 days)
Change from Baseline in Macrophages Cell Count for Q3W Schedule | PrI (0 hr) on Cy1D1 (Baseline), Cy1 Day 21, and Cy3 Day 21 (Cycle length = 21 days)
Change from Baseline in Cytokines Level for Q2W Schedule | PrI (0 hr) on Cy1D1 (Baseline), Cy1 Day 14, and Cy4 Day 14 (Cycle length = 14 days)
Change from Baseline in Cytokines Level for Q3W Schedule | PrI (0 hr) on Cy1D1 (Baseline), Cy1 Day 21, and Cy3 Day 21 (Cycle length = 21 days)
Change from Baseline in HER3 Expression for Q2W Schedule | PrI (0 hr) on Cy1D1 (Baseline), Cy1 Day 14, and Cy4 Day 14 (Cycle length = 14 days)
Change from Baseline in HER3 Expression for Q3W Schedule | PrI (0 hr) on Cy1D1 (Baseline), Cy1 Day 21, and Cy3 Day 21 (Cycle length = 21 days)
Change from Baseline in Phosphorylated HER3 Expression for Q2W Schedule | PrI (0 hr) on Cy1D1 (Baseline), Cy1 Day 14, and Cy4 Day 14 (Cycle length = 14 days)
Change from Baseline in Phosphorylated HER3 Expression for Q3W Schedule | PrI (0 hr) on Cy1D1 (Baseline), Cy1 Day 21, and Cy3 Day 21 (Cycle length = 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- Rigshospitalet, Onkologisk Klinik, København Ø, Denmark
- Netherlands (4):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Academ Ziekenhuis Groningen; Medical Oncology, Groningen
  - Erasmus Medisch Centrum Rotterdam; Lokatie Daniel den Hoed, Rotterdam
  - Utrecht University Medical Centre; Dept of Medical Oncology and UPC, Utrecht
- South Korea (2):
  - National Cancer Center, Gyeonggi-do
  - Asan Medical Center, Seoul
- Spain (5):
  - Hospital del Mar; Servicio de Oncologia, Barcelona, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona, Barcelona
  - Centro Integral Oncologico Clara Campal (CIOCC); Dirección Médica, Madrid, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville, Sevilla
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia, Valencia

REFERENCES:
- [Derived] Kim HS, Han JY, Shin DH, Lim KY, Lee GK, Kim JY, Jacob W, Ceppi M, Weisser M, James I. EGFR and HER3 signaling blockade in invasive mucinous lung adenocarcinoma harboring an NRG1 fusion. Lung Cancer. 2018 Oct;124:71-75. doi: 10.1016/j.lungcan.2018.07.026. Epub 2018 Jul 20. PMID 30268483